CLINICAL TRIAL: NCT04649294
Title: The Effect of High Dose Glucocorticoid Steroids on Myocardial Function
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0052-17
Record Dates: First submitted 2020-10-24; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-10

CONDITIONS: High-dose Steroids, Myocardial Function, Longitudinal Strain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long term steroid exposure, as in Cushing's disease, causes myocardial dysfunction, hypertrophy and fibrosis in addition to causing obesity, hypertension and glucose intolerance. The aim of our study was to verify if short-term high-dose exogenous steroid therapy adversely effects the heart.

DETAILED DESCRIPTION:
Patients eligible for high dose steroid therapy due to inflammatory diseases were offered to participate in this study. The minimal total intravenous dose was 375 mg prednisone, and the daily steroids were divided into 2-3 doses. To determine the steroids' effect on myocardial function the echocardiographic studies included estimation of global and segmental longitudinal strain. Each patient had a baseline echocardiographic study performed before high-dose steroid therapy was initiated and again immediately after it. A follow-up echo study was performed after completion of a 3-month low-dose steroid therapy period. The paired 2-tailed t-test was used to compare group means

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Patient with rheumatic disease that need high dose steroids due to exacerbation
* Patient whom echocardiographic study can be performed with a good quality

Exclusion Criteria:

* age below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with inflammatory disease who needs high dose steroids according to there disease severity and welling to participate in observation study to see the effect od steroids taken on the myocaridal functions duering hospital stay
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
determine the steroids' effect on myocardial function the echocardiographic studies included estimation of global and segmental longitudinal strain | two years
  the aim of the study was to verify if the reported adverse effect of long-term endogenous cortisol excess on LV systolic and diastolic function occurs after short-term, high-dose, exogenous steroid therapy as well.Patients with inflammatory diseases in internal medicine department who needed treatment with high dose steroids recruited to the study baseline echocardiographic study performed before high-dose steroid therapy was initiated. A second study was performed after completion of the high-dose protocol and scheduled for a third echocardiographic study after completion of a 3-month low-dose steroid therapy period or immediately after termination of steroid therapy if it was during the 3-month period . global and segmental longitudinal strain measured by echo in addition to standard echo measures .the aim to see if high dose steroids use accompanied by echocardiographic changes as seen in Cushing disease

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Hospital, Hadera, Israel